CLINICAL TRIAL: NCT06949644
Title: Pupillometry in DSWPD Type 1 and Type 2
Brief Title: Pupillometry in Delayed Sleep Wake Phase Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sabra Abbott, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00221304; R01HL174661 (NIH)
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Delayed Sleep-Wake Phase Disorder
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — Light; Citalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DSWPD (Experimental): Placebo or Citalopram followed by bright light (all participants will receive both interventions in random order).
  Interventions: Combination Product: Light and Citalopram

INTERVENTIONS:
Combination Product: Light and Citalopram — Participants will receive placebo or citalopram, followed by bright light exposure

SUMMARY:
The goal of this observational study is to characterize the pupil light response in patients with delayed sleep-wake phase disorder. A subset of participants will take part in a clinical trial to determine if increasing serotonin can alter the circadian response to light. The main questions it aims to answer is:

Are there differences in the light response in patients with delayed sleep-wake phase disorder? Does citalopram increase melatonin suppression in patients with delayed sleep-wake phase disorder?

Participants will complete activity and melatonin testing at home to determine their circadian timing. This will be followed by an eye test looking at the pupil response to different light stimuli. A subset of participants will complete two inpatient admissions where melatonin levels will be sampled and they will be exposed to a bright light. During one round of testing they will receive a placebo and in the other round of testing they will take a single dose of citalopram, a selective serotonin reuptake inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Delayed sleep-wake phase disorder

Exclusion Criteria:

* Use of medications known to alter pupil diameter
* History of eye disease or eye surgery
* Unstable medical or psychiatric condition
* Shift work or self imposed irregular sleep schedules
* Caffeine consumption >400mg/day

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Melatonin suppression | 8 hours
  Saliva melatonin samples will be collected before and after light exposure

IPD SHARING:
Plan to Share IPD: Undecided